CLINICAL TRIAL: NCT00472550
Title: Effects of Esomeprazole on Gastric Emptying of Alcoholic Beverages, Blood Alcohol Concentrations, Gastroesophageal Reflux and Release of Some Gastrointestinal Hormones in Healthy Volunteers
Brief Title: Esomeprazole and Gastric Emptying of Beer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Mannheim-Eso-001
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2007-05-11 (Estimated); Status verified 2007-05

CONDITIONS: Gastroesophageal Reflux; Heartburn
Keywords: esomeprazole, gastric emptying, reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: esomeprazole 20 mg

SUMMARY:
To investigate the effect of 20 mg esomeprazole daily for one week on gastric emptying of 500 ml beer, the consecutive blood alcohol levels, the gastroesophageal reflux and plasma levels of gastrin and CCK in a randomized, placebo-controlled, double-blinded manner in 16 healthy male volunteers.

Hypothesis:

The combined taking of esomeprazole and beer will inhibit gastric emptying as compared to the intake of beer alone. This will induce a delay of the ethanol absorption and of the consecutive blood ethanol concentrations. Gastric acid secretion after beer will be reduced after esomeprazole treatment. Therefore, gastroesophageal acid reflux will be reduced after the combined taking. We speculate that gastrin, but not CCK plasma levels, will be increased after the combined taking as compared to beer alone. Both, beer and PPIs, have stimulatory effects on gastrin release. However, the secretion of CCK from duodenal CCK-cells is inhibited when gastric emptying is prolonged.

DETAILED DESCRIPTION:
Sixteen healthy, male and non-smoking volunteers will be enrolled in this study. The subjects will be treated with placebo or with 20 mg esomeprazole daily for one week before gastric emptying will be determined. The sequence of the tests (verum or placebo) will be randomised in a cross over design. In each subject at most one test will be performed every 2 weeks to ensure one week without treatment (wash-out-phase) between both experiments.

All examinations will be performed in the afternoon. After a small breakfast in the morning subjects fast for at least 8 hours. During the examination, all subjects are sitting slightly leaned backwards. A double lumen nasogastric tube (Ch 14, Laboratories Pharmaceutiques Vygon, Ecouen, France) will be positioned in the most dependent part of the stomach and a pH-probe (F8/IR blue line, SME Medizintechnik, Weil am Rhein) will be positioned 5 cm above the lower esophageal sphincter. 500 ml beer will then be instilled into the stomach over 5 min. Gastric emptying will be determined every 10 min for 2 hours by ultrasonography.

Withdrawal criteria The trial can be stopped anytime by the volunteer without specified reasons or by the investigator in case of incompliance of the volunteer or subsequent incidence of exclusion criteria. In case of hypersensitive or allergic reaction against the medication or side effects of the medication, such as urtication, angioneurotic edema, vomiting, cardiovascular reaction (systolic blood pressure under 100 mm/Hg), paraesthesia, confusion, bronchial spasm or fever, the study will also be stopped.

In case of withdrawal of volunteers, up to four additional volunteers can be recruited to complete totalling 16 volunteers.

Assessment of safety Esomeprazole is a frequently administered drug in the therapy of particularly gastroesophageal reflux disease, gastritis and gastric or duodenal ulcers. Side effects are very rare, headache, abdominal pain, diarrhoea, bloating, nausea, vomiting and constipation are thereof the most frequent. The methods used in this study are clinical routine procedures and imply -if used by skilful physicians as in this study - no risk for complications.

To detect side effects or complications the investigator is present in the examination room during the whole study and blood pressure and heart rate are measured every 15 minutes. Before the each study and during the introduction procedure a physical examination will be performed by the investigator.

Ultrasonography Ultrasonography of the antrum and the fundus represents a highly reliable and reproducible radiation-avoiding method for determination of gastric emptying [11-14]. To determine gastric emptying of the proximal and distal stomach, we will use a curved array scanner with a 3.25 MHz ultrasound transducer (Sonoline Sienna®; Siemens, Germany). We determine emptying of the distal stomach by measuring the cross-sectional area of the antrum at the level of the superior mesenteric vein and the aorta [12, 13]. The vessels are used to standardize the position of the scans. This antral area is scanned before, immediately after intragastrical application of the test solution and every 10 minutes for two hours.

Gastic emptying of the proximal stomach will be measured immediately after the application and every 10 min until the fundus is emptied completely using the following ultrasonographic method: the transducer will be positioned in the epigastrium at the left subcostal margin and tilted cranially. The maximal angle of view of the scanner is used to visualize as much of the proximal stomach as possible. Two standardized sonographic image sections are chosen: First, a sagital section with the left renal pelvis in a longitudinal projection, the left lobe of the liver and the tail of the pancreas as internal landmarks. The transducer is then rotated 90° clockwise to obtain an oblique frontal section where the left hemidiaphragm, the top margin of the fundus, and the liver parenchyma serve as landmarks. A proximal gastric area is outlined in the sagital section by tracing from the top margin of the fundus and 7 cm downward along the axis of the stomach. The maximal diameter in the oblique frontal section, kept within 7 cm along the axis of the proximal stomach, is chosen as the second measure. Both measurements are combined to estimate an approximate volume of the fundus [11].

The inner echogenic layer corresponding to the interface between the gastric content and the mucosa of the gastric wall is outlined. The measurements were repeated twice and the mean value is used. The areas of the antrum and the fundus and the diameter of the fundus are traced by the internal calliper provided with the ultrasound instrument. All ultrasonographic parameters will be measured twice, the mean of both measurements will be chosen to be representative.

Gastric half emptying time (t(1/2)) will determined separately for the fundus and the antrum.

Plasma gastrin, plasma CCK and serum ethanol concentrations Blood samples (10 ml) will be drawn at baseline and every 15 min after application of the test solution for 2 hours for the determination of serum ethanol concentrations. Samples will be centrifuged immediately at 4° C. The serum concentration of ethanol will be determined using the alcohol-dehydrogenase method (Ethylalkohol, Roche Diagnostics GmbH, Mannheim, Germany). The plasma concentrations of gastrin will be measured by the Institute for Clinical Chemistry at the University Hospital Mannheim by radioimmunassays (RIA) and that of CCK at the Universityhospital Basel (Professor Ch. Beglinger, no round robin test certificate available).

Gastroesophageal reflux The intraesophageal pH (5 cm above the lower esophageal sphincter) will be recorded for 4 hours by GastroScan II (SME Medizintechnik, Sprendlingen). The correct position of the tip of the pH-probe will be measured by pH-metry during the visit for the screening examinations. The portion of intraesophageal pH<4 and the DeMeester-Score (frequency and duration of pH<4) will be calculated.

Gastrointestinal complaints The volunteers mark additionally on a visual analogue scale (VAS 0-100) their intensity of fullness, bloating, heartburn and satiety before the ingestion of beer and than in 10 min intervals for 2 hours.

Statistical analysis Statistical significances for differences between gastric emptying rates, blood alcohol concentrations and gastroesophageal reflux will be determined using student´s t-test.

ELIGIBILITY:
Inclusion Criteria:

* Male, non-smoking volunteers without regular medication or regular alcohol consumption will be included.
* Before inclusion blood will be drawn and the following blood count, liver, pancreas, kidney, thyroid and coagulation parameters will be examined:

  * Creatinine (0.5 - 1.3 mg/dl),
  * Alc. Phosphatase (38 - 126 U/l),
  * GGT (0 - 85 U/l),
  * ALAT (0 - 50 U/l),
  * ASAT (0 - 37 U/l),
  * LDH (0 - 248 U/l),
  * Cholinesterase (>7000 U/l),
  * Amylase (25 - 130 U/l),
  * Lipase (114 - 300 U/l),
  * Leucocytes (3,5 - 11.0 10E9/L),
  * Erythrocytes (4.0 - 5.9 10E12/L),
  * Hb (12.0 - 17.5 g/dl),
  * Ht (33 - 50%),
  * Platelets (145 - 440 10E9/L),
  * CrP (< 10 mg/l),
  * TSH (0.4 - 5.0 mE/l),
  * fT4 (6 - 23 pmol/l),
  * INR (0.75 - 1.30),
  * PTT (15.0 - 33.0 sec.)

The results have to be within the physiological range (as given in parenthesis).

Moreover, volunteers have mentally to be able to understand the explanations concerning the study and follow to the instructions of the investigator.

Exclusion Criteria:

* Any acute or chronic disease,
* Heartburn more than once weekly,
* Alcohol consumption of more than 50 g ethanol-equivalent per week,
* Smoking,
* Known hypersensitivity against esomeprazole,
* Benzimidazole or other ingredients of the medication,
* Fructose-intolerance,
* Glucose-galactose-malabsorption or saccharase-isomaltase-deficiency.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-01; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Gastric emptying time, gastroesophageal reflux | 3h

SECONDARY OUTCOMES:
blood ethanol concentration, CCK-levels, gastrin-levels, dyspeptic symptoms | 3h

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Franke, MD, Principal Investigator — Dep. Medicine II, University hospital Mannheim
Locations (1):
- Dep. Medicine II, University Hospital Mannheim, Mannheim, Germany